CLINICAL TRIAL: NCT01471197
Title: A Randomized, Open-Label, Phase 2 Safety and Efficacy Trial of Ipilimumab Versus Pemetrexed in Subjects With Recurrent/Stage IV Non-Squamous, Non-Small Cell Lung Cancer Who Have Not Progressed After Four Cycles of a Platinum-Based First Line Chemotherapy
Brief Title: Safety and Efficacy Trial of Ipilimumab Versus Pemetrexed in Non-Squamous Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-124 ST; 2011-000732-29 (EudraCT Number)
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Lung Cancer - Non Small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Ipilimumab (Experimental)
  Interventions: Biological: Ipilimumab
- Arm 2: Pemetrexed (Active Comparator)
  Interventions: Biological: Pemetrexed

INTERVENTIONS:
Biological: Ipilimumab — Intravenous (IV) solution, IV, 10mg/kg, Once every 3 weeks for 4 doses, then once every 12 weeks during Treatment Phase, 90 minute infusion
  Other Names: Yervoy; BMS-734016
  Arms: Arm 1: Ipilimumab
Biological: Pemetrexed — IV solution, IV, 500 mg/m2, Once every 3 weeks during Treatment Phase, 10 minute infusion.
  Other Names: Alimta
  Arms: Arm 2: Pemetrexed

SUMMARY:
The purpose of this trial is to determine whether Ipilimumab will prolong survival when compared to Pemetrexed in subjects with nonsquamous, non-small cell lung cancer.

ELIGIBILITY:
For additional information, please contact the BMS oncology clinical trial information service at 855-216-0126 or email MyCancerStudyConnect@emergingmed.com. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Inclusion Criteria:

* Non-Squamous, Non-Small Cell Lung Cancer
* Recurrent/Stage IV Non-small cell lung cancer (NSCLC)
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Not progressing after 4 cycles of a platinum-based first line chemotherapy

Exclusion Criteria:

* Brain Metastases (unless stable)
* Autoimmune Diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- United States (7):
  - Marin Specialty Care, Inc., Greenbrae, California
  - Medical And Surgical Specialists, Llc, Galesburg, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - Meritus Center For Clinical Research, Hagerstown, Maryland
  - Carolina Biooncology Institute, Huntersville, North Carolina
  - Blue Ridge Cancer Care, Christiansburg, Virginia
- Belgium (2):
  - Local Institution, Bruges
  - Local Institution, Sint-Niklaas
- Local Institution, Paris, France
- Germany (2):
  - Local Institution, Hamburg
  - Local Institution, Heidelberg
- Local Institution, Benidorm-Alicante, Spain

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started July 2012 and completed February 2013. After 9 participants enrolled, the study was terminated for administrative reasons unrelated to adverse events (AEs) or expectation of efficacy associated with either ipilimumab or pemetrexed.
Pre-assignment Details: 9 participants enrolled; 8 participants randomized; 1 participant not randomized due to disease progression and death.
Groups:
- Ipilimumab 10 mg/kg: Ipilimumab: Intravenous (IV) solution, IV, 10 milligrams per kilogram (mg/kg), Once every 3 weeks for 4 doses, then once every 12 weeks during Treatment Phase, 90 minute infusion.
- Pemetrexed 500 mg/m^2: Pemetrexed: IV solution, IV, 500 milligram per meter squared (mg/m^2), Once every 3 weeks during Treatment Phase, 10 minute infusion.
Period: Overall Study
Arm/Group | Ipilimumab 10 mg/kg | Pemetrexed 500 mg/m^2
Started | 6 | 2
Completed | 0 | 0
Not Completed | 6 | 2
Not completed — Disease Progression | 4 | 2
Not completed — Death | 1 | 0
Not completed — Study Drug Toxicity | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least one dose of either study medication.
Groups:
- Pemetrexed 500 mg/m^2: Pemetrexed: IV solution, IV, 500 mg/m^2, Once every 3 weeks during Treatment Phase, 10 minute infusion.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab 10 mg/kg | Pemetrexed 500 mg/m^2 | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.85) | 61.0 (1.41) | 62.3 (7.54)
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 4 | 2 | 6
  Greater than, equal to (>=) 65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 1 | 5
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group Performance Status (ECOG PS) is a questionnaire which measures the activity of a an oncology patient. Measurements range from 0 to 5 with 0=fully active; 1= restricted in physically strenuous activity; 2= ambulatory; 3=limited self care; 4= completely disabled; 5=dead.
  participants
    ECOG PS 0 | 3 | 1 | 4
    ECOG PS 1 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival of Participants During the Study - All Treated Participants
Description: Overall survival (OS) was defined as the time from the date of randomization until the date of death. For those participants who did not die by the time the study was terminated and last patient, last visit occurred, OS was censored (+) on the last date the participant was known to be alive. OS is presented below in increasing monthly categories of survival. OS analysis was to be performed when a total of approximately 132 deaths were observed but due to the early termination of the study, statistical analyses were not performed.
Time Frame: Date of Randomization to date of death, up to last patient, last visit, approximately 7 months after study started
Population: All participants who received at least one dose of either study drug.
Measure: Number; unit: participants
Arm/Group | Ipilimumab 10 mg/kg | Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 6 | 2
participants
  Overall Survival 0.9 months | 1 | 0
  Overall Survival 1.8 months | 1 | 0
  Overall Survival 3.9 months+(censored) | 1 | 0
  Overall Survival 4.4 months+(censored) | 2 | 0
  Overall Survival 4.6 months+(censored) | 1 | 0
  Overall Survival 5.4 months+(censored) | 0 | 2

2. Secondary Outcome: Number of Participants Who Died Within 30 Days and 31 Days After Last Dose - All Treated Participants
Description: Due to study termination, the categories presented below are deaths occurring within 30 days of last dose and deaths occurring within 32 days of last dose. If the study had not been terminated early, the categories presented would have been 30 days and 90 days after last dose.
Time Frame: Day 1 of Treatment to Date of Death, up to last patient, last visit, approximately 7 months after study started.
Population: All participants who were randomized and treated with at least one dose of either study drug.
Measure: Number; unit: participants
Arm/Group | Ipilimumab 10 mg/kg | Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 6 | 2
participants
  Death within 30 Days of Last Dose | 1 | 0
  Death within 32 Days of Last Dose | 1 | 0

3. Secondary Outcome: Number of Participants With Deaths, Adverse Events (AEs), Serious AEs (SAEs) and AEs Leading to Discontinuation - All Treated Participants
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling. Participants were evaluated from Day 1 (first day of treatment with study drug) to the date of the last participant, last visit of the study.
Time Frame: Day 1 to Date of last patient, last visit, approximately 7 months after study started.
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ipilimumab 10 mg/kg | Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 6 | 2
participants
  Deaths | 2 | 0
  SAEs | 5 | 1
  AEs | 6 | 2
  AEs leading to discontinuation | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Last patient, last visit, approximately 7 months after start of study.
Description: Study initiated 11 July 2012, was terminated and last patient, last visit was 25 Feb 2013
Arm/Group | Ipilimumab 10 mg/kg | Pemetrexed 500 mg/m^2
Serious Adverse Events (participants affected / at risk) | 5/6 | 1/2
Other Adverse Events (participants affected / at risk) | 5/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab 10 mg/kg (N=6) | Pemetrexed 500 mg/m^2 (N=2)
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab 10 mg/kg (N=6) | Pemetrexed 500 mg/m^2 (N=2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Amylase increased (Investigations) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0

LIMITATIONS AND CAVEATS:
At the time of the early termination of this study, most participants only had only one on-study tumor assessment performed. Therefore, the tumor response-related endpoints were too immature to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.